CLINICAL TRIAL: NCT03891589
Title: Promotion of Optimized Complementary Feeding With or Without Home Fortification (Taburia) Prevents the Decrease of Nutrient Intake, Level of Micronutrient, and Anthropometric Indices, Also Digestive Health Among Under-Five Children
Brief Title: Optimized Complementary Feeding With or Without Home Fortification Prevents Decrease of Micronutrient and Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Kadek Tresna Adhi, Principal Investigator, Udayana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UdayanaU_01
Record Dates: First submitted 2019-03-14; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Complementary Feeding; Linear Programming; Nutritional Status; Micronutrient Deficiency; Growth Failure
Keywords: Complementary feeding; Linear Programming; Nutritional status; Micronutrient; Growth
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Intervention Model Description: The intervention groups consisted of promotion of optimized complementary feeding (CF) with taburia (P1, n=51), optimized CF (P2, n=54) and taburia home fortification (P3, n=47). Control groups will not receive intervention or placebo but will receive only a standardized primary health care education program related to complementary feeding practices for infants and children. Also, the nutritional status of all groups will be measured every month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Optimized CF with Taburia (Experimental): The intervention groups consisted of promotion of optimized complementary feeding with home fortification (taburia) one sachet per week
  Interventions: Behavioral: Nutritional education program; Dietary Supplement: Home fortification (Taburia)
- Optimized CF only (Experimental): The intervention groups consisted of promotion of optimized complementary feeding without home fortification (taburia)
  Interventions: Behavioral: Nutritional education program
- Taburia (Experimental): The intervention groups consisted of provision taburia home fortification three sachet per week
  Interventions: Dietary Supplement: Home fortification (Taburia)
- Control (No Intervention): No intervention but gave a standard education from primary health center

INTERVENTIONS:
Behavioral: Nutritional education program — These programs were a process of providing information or knowledge to mother of the children consisting of information on initiation of complementary feeding, variety, and frequency of food, nutrient requirements and diet pattern for children (the amount and types of food), and benefits of Taburia. All this information provided through class-based activities and group discussion by using leaflet and food model conducted by the researchers. Education materials developed based on CFR models from our previous study by applying the LP approach. There was also a demonstration on administering complementary feeding (demo and cooking class) to improve skills of the mother on food from selection, design, handling and preparing, based on requirements of the children. This activity conducted through training once per month for the first four months of the intervention. Components of complementary feeding promoted in this study are based on CFR using LP approach from our previous research.
  Arms: Optimized CF only; Optimized CF with Taburia
Dietary Supplement: Home fortification (Taburia) — Taburia is a multivitamin and mineral fortification to provide sufficient amount of nutrient for optimal growth and development of children aged 6-59 months. Every sachet of Taburia prepared to fulfill minimum nutrient requirements for children aged 6-59 months. Each sachet is one gram in weight and contains vitamin A (417 mcg), B1 (0.5 mg), B2 (0.5 mg), B3 (5.0 mg), B6 (0.5 mg), B12 (1 mcg), D3 (5 mcg), E (6 mg), K (20 mcg), C (30 mcg), folic acid (150 mcg), pantothenic acid (3 mcg), Iodium (50 mcg), Iron (10 mg), Zn (5 mg) and Selenium (20 mcg). One sachet of Taburia given to the subject by adding it to their breakfast and must be finished. The frequency of Taburia consumption per week follows the finding of the LP analysis from the previous study. Taburia intervention complemented by health education related to benefits, administration of Taburia, and its side effects. Compliance will be evaluated directly by the researcher based on empty Taburia sachet and conducted every month.
  Arms: Optimized CF with Taburia; Taburia

SUMMARY:
Malnourished among under-five children characterized by growth faltering is a public health concern in Indonesia. It requires serious action from the governments because of the prevalence of underweight, stunting, and wasting are increasing. These impacts are irreversible resulting in the low quality of future human resources. Several studies showed that growth faltering among under-five children starts at age six months when the amount of breastmilk reduced, complementary feeding initiated, and risk for infection is increased. A rapid growth phase also causes growth faltering at age 6-24 months. The inadequate amount and low quality of food during this period can also lead to reducing nutritional status. The Indonesian Government released a national policy in 2013 to address undernutrition among under-five children called the Indonesia President Regulation No. 42/2013 regarding national movements on the acceleration of nutritional programs to address micronutrients deficiency among under-five children by providing micronutrient powder (MNP) (called Taburia) for children aged 6 - 59 months. Our literature review documented that there is no study ever conducted to evaluate the effectiveness of MNP (Taburia) in improving the weight and height of the children. Moreover, behavioral modification interventions to promote food diversification to improve nutrient intake and to prevent micronutrient deficiency are also never conducted. Based on the rationale and study concept, the following hypotheses are 1). Promotion of optimized complementary feeding along with or without multi-micronutrient powder or MNP (namely taburia) can prevent reductions in nutrient intake and density; serum ferritin and zinc levels; and anthropometric z-score index compared to controls, and 2) provision of MNP can prevent reductions in nutrient intake and density; serum ferritin and zinc levels; and anthropometric z-score index compared to controls.

DETAILED DESCRIPTION:
Our study consists of two phases. The first phase was to develop a combination model of Complementary Feeding Recommendation (CFR) or optimized Complementary Feeding (CF) with or without MNP home fortification (Taburia) by using a Linear Programming approach. The objective of this stage was to address the nutrient gaps. Also, nutrient analysis of Taburia by employing an LP approach will provide adequate dosing of Taburia to added to local CF. Several studies have documented that MNP supplementation associated with a reduced bacterial population in digestive systems (Lactobacillus dan Bifidobacterium spp) and induced inflammation on the intestines. These conditions reduce the absorption capacity of digestive systems leading to nutrient deficiency among under-five children. Findings from the first phase were an optimized model of CF with or without MNP (Taburia) as an intervention media in the second phase of our study, which evaluates the effectiveness of a combination of CFRs and MNP fortification using an LP approach. This intervention group compared to (1) optimal Complementary Feeding (CF) with MNP one sachet per week, (2) optimized CF group alone, (3) Provision MNP alone three sachets per week, and (4) control group. Several indicators to be evaluated were (1) nutrient intake and density; (2) z-score of anthropometric index; (3) micronutrient status; (4) digestive health status (relative population of DNA Bifidobacterium and Lactobacillus spp).

ELIGIBILITY:
Inclusion Criteria:

* Under-five children aged 6-11 months (baseline) with normal nutritional status based on weight for height/length z-score (more than -2 SD based on the World Health Organization (WHO) Growth standard (2006))
* Resided in the study location
* Parent or carer agreed to participate in the study and have signed informed consent.

Exclusion Criteria:

* Children with poor nutritional status (<-2SD based on WHZ)
* Families refusing to participate

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline nutrient intake at 6 months | Before intervention and after six month periode intervention
  Data related to nutrient intake nutrient before and after the intervention measured using a 24-hour recall and a food frequency questionnaire and collected through a structured interview. Also, data related to compliance, side effects, and acceptability of MNP home fortification (Taburia) evaluated directly by the research team during the intervention period. Nutrient composition in-home fortification (Taburia) also includes in analysis Nutrisurvey software.
Change from baseline nutrient density at 6 months | Before intervention and after six month periode intervention
  Data related to nutrient density before and after the intervention measured using a 24-hour recall and a food frequency questionnaire and collected through a structured interview. Nutrient density is calculated from intake ratio or total nutrient obtained from the diet divided by total energy from the diet per 100 kcal. Dietary data measured using a food scale (Tanita KD-160) as well as household measurements such as glass, plate, spoon, bowl, and others.
Change from baseline level of serum ferritin at 6 months | Before intervention and after six month period intervention
  Serum ferritin level measured by the Enzyme-linked immunosorbent assay (ELISA) kit (Bioassay Technology Laboratory) Cat. No. E1702Hu and expressed in units of μg/ml.
Change from baseline Level of zinc serum at 6 months | Before intervention and after six month period intervention
  The serum zinc level measured using the GBC 933 AA type atomic absorption spectrophotometer (AAS) with a wavelength of 213.9 nm and expressed in units of μmol/L.
Change from baseline z-score anthropometry indices at 6 months | Carried out routinely every month for six months, starting at the beginning before and at the end of the intervention.
  Weight and height of the children measured before the intervention and will be followed by regular measurement every month until the end of the intervention period. These data analyzed using the WHO Anthro 2005 software to calculate z-score anthropometric index (weight for age, length for age, weight for height) and presented as z-score to determine the nutritional status of our samples. Body weight measured using a digital EBSC infant weigher with the accuracy of 0.01 kg and using a standing digital weigher (CAMRY) with an accuracy of 0.01 kg for children who already can stand up. Length or height measured using a length board (SECA 210) with an accuracy of 0.01 cm.

SECONDARY OUTCOMES:
Hemoglobin level | Measured at the end or after six month period of intervention
  Hemoglobin level was carried out to determine the anemia status in children under five with the Flowcytometry method expressed in g/dL.
Change from baseline infection status (hs-CRP level) at 6 month | Before intervention and after six month period intervention
  The hs-CRP level is an examination to measure the concentration of C-reactive protein which is more sensitive, measured by the enzyme-linked immunosorbent assay (ELISA) kit (Bioassay Technology Laboratory) Cat. No. E1805Hu and expressed in mg/L units.
Gut microbiota | Measured at the end or after six month period of intervention
  The relative proportion of digestive tract bacterial DNA is the relative proportion of the DNA population of Bifidobacterium and Lactobacillus spp bacteria compared to the controls analysed using the qPCR method.
Helminth status | Measured at the end or after six month period of intervention
  The helminthiasis was carried out using the Kato-Katz method
Dietary diversity | After six month period of intervention
  The food diversity score is calculated by summing the number of food groups consumed by individual respondents during the 24-hour recall period. Scoring is done by giving a score of one if consuming and a score of 0 if not consuming one type of food contained in a food group that has been determined by FAO.
Adherence to home fortification (taburia) | Carried out routinely every month for six months until the end of the intervention.
  Adherence with the provision of taburia is the adherence of the mother or caregiver in giving taburia to the subject during the intervention program and is monitored directly by the researcher and field worker by collecting the number of sachets spent each month. The provision of taburia is given once a month as many as four sachets for group optimized CF with taburia and 12 sachets for group taburia only.

CONTACTS AND LOCATIONS:
Overall Officials: Kadek T Adhi, Principal Investigator — Udayana University
Locations (1):
- Susut District, Bangli, Bali, Indonesia